CLINICAL TRIAL: NCT04572191
Title: Ceramide Level as Apredictor of Outcomes in Patients of Anterior Myocardial Infarction Undergoing Primary Coronary Intervention
Acronym: STEMI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, esraa sayed hamed Ahmed, principle investigator, Assiut University
Other Study IDs: anterior STEMI
Record Dates: First submitted 2020-09-27; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Anterior STEMI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CERAMIDE LEVEL IN BLOOD — BY ELISA ASSAY TO DETECT CERAMIDE LEVEL IN BLOOD IN ANTERIOR STEMI PATIENTS

SUMMARY:
Ceramide level as a predictor of outcomes in patients of anterior myocardial infarction undergoing primary Coronary intervention

DETAILED DESCRIPTION:
Ceramides are a family of lipid molecules that are found in high concentrations within cell membranes and play a key role in a variety of physiological functions including apoptosis, cell growth, cell adhesion and plasma membrane integrity maintenance.(1)

All tissues can synthesize ceramides de novo from saturated fats and sphingosine.(2) the ( LDL ) Present in atherosclerotic plaque is rich in ceramide and contain 10 - 50 fold higher content of ceramide when compared with plasma LDL .(3)

Ceramide (d18:1/16:0) is associated with the fraction of necrotic core tissue and lipid core burden in coronary atherosclerosis.(4) Previous clinical research found that circulating ceramides are elevated in patients with hypertension,(5) obesity (6 - 7) and type II diabetes mellitus.

Previous clinical research found that elevated ceramide plasma concentrations are associated with coronary plaque vulnerability evaluated by intravascular ultrasound .

virtual Recent studies showed targeted profiling of ceramides predicted short-term and long-term major adverse cardiac events.

Plasma ceramide level is also positively associated with the levels of total cholesterol. [8 - 9] The plasma ceramides that have been studied as high-risk factors are Cer (d18:1/16:0), Cer (d18:1/18:0) and Cer (d18:1/24:1) and the ratios of these ceramides to Cer (d18:1/24:0) [10 - 11].

However, it is tempting to speculate that ceramides are associated with plaque vulnerability as they are known to fuel many central atherosclerosis processes including lipoprotein aggregation and uptake, inflammation, superoxide anion production, andapoptosis 12 - 13 - 14

ELIGIBILITY:
Inclusion Criteria:

* 1- Subjects with anterior STEMI according to ESC guidelines 2017 . 2. Subjects undergoing PPCI

Exclusion Criteria:

* Patients with previous PCI. Patients with previous CABG. Patients with TIMI flow less than II. Patients with residual stenosis more than 70 % in major artery. Cardiogenic shock.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALL PATIENTS COMPLAING OF ANTERIOR STEMI & UNDERENTPRIMARY PCI
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
to detect early & mid -term MACE complication in anterior STEMI patients undergoing PPCI & their relation with ceramide level in these patients | BASELINE
  to detect early & mid -term MACE complication in anterior STEMI patients undergoing PPCI & their relation with ceramide level in these patients

CONTACTS AND LOCATIONS:
Overall Officials: mohamed abdel - ghani, professor, Principal Investigator — Assiut University
Locations (1):
- Esraa Sayed Hamed, Asyut, Egypt

REFERENCES:
- [Background] Tu C, Xie L, Wang Z, Zhang L, Wu H, Ni W, Li C, Li L, Zeng Y. Association between ceramides and coronary artery stenosis in patients with coronary artery disease. Lipids Health Dis. 2020 Jun 25;19(1):151. doi: 10.1186/s12944-020-01329-0. PMID 32586390
- [Background] Pan W, Li L, Sun M, Wang C, Fang S, Yu B. Plasma ceramides are associated with coronary atherosclerotic burden in patients with ST-segment elevation myocardial infarction. Int J Cardiol. 2020 Dec 1;320:155-160. doi: 10.1016/j.ijcard.2020.08.010. Epub 2020 Aug 12. PMID 32800902
- [Background] Mantovani A, Bonapace S, Lunardi G, Canali G, Dugo C, Vinco G, Calabria S, Barbieri E, Laaksonen R, Bonnet F, Byrne CD, Targher G. Associations between specific plasma ceramides and severity of coronary-artery stenosis assessed by coronary angiography. Diabetes Metab. 2020 Apr;46(2):150-157. doi: 10.1016/j.diabet.2019.07.006. Epub 2019 Aug 3. PMID 31386900
- [Background] Tu CC, Wan BY, Zhao XL, Li CX, Wu HM, Zhang LL, Li L, Zeng Y. [Value of ceramide in the diagnosis and risk prediction of coronary artery disease]. Zhonghua Yi Xue Za Zhi. 2019 Oct 22;99(39):3089-3092. doi: 10.3760/cma.j.issn.0376-2491.2019.39.010. Chinese. PMID 31648453